CLINICAL TRIAL: NCT00571454
Title: Culturally Sensitive Depression Care Management for Latino Primary Care Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Neighborhood health Plan of RI (Unknown); Beacon Health Strategies (Industry); Robert Wood Johnson Foundation (Other)
Responsible Party: Beth Marootian, Director of Business Development, Neighborhood Health Plan of RI
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RWJ
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Depression
Keywords: depression; primary care; Latino; telephone; care management
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Telephone depression care management + treatment as usual
  Interventions: Behavioral: telephone depression care management
- 2 (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: telephone depression care management — 1 call per week for first 4 weeks
  1 call every other week for next 8 weeks
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether telephonic depression care management can improve depression outcomes for Latino primary care patients who are enrolled in Medicaid and are receiving an antidepressant from their primary care doctor.

ELIGIBILITY:
Inclusion Criteria:

* Latino
* Adult
* Received an antidepressant prescription from primary care provider
* Not current receiving care from behavioral health provider
* Diagnosis of major depression, minor depression, dysthymia, or significant depression symptoms
* English or Spanish speaking
* Member, Neighborhood Health Plan of RI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Clinician Administered (QIDS-C) | 3 months

SECONDARY OUTCOMES:
Center for Epidemiological Studies-- Depression | 3 months
WHO Disability Assessment Schedule (WHO-DAS) | 3 months
Treatment Utilization | 3 months
Treatment Satisfaction | 3 months
costs: health care utilization | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth Ann Marootian, MPH, Principal Investigator — Neighborhood health Plan of RI; Ivan W Miller, PhD, Principal Investigator — Butler Hospital; Lisa A Uebelacker, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Neighborhood Health Plan of RI, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Uebelacker LA, Marootian BA, Tigue P, Haggarty R, Primack JM, Miller IW. Telephone depression care management for Latino Medicaid health plan members: a pilot randomized controlled trial. J Nerv Ment Dis. 2011 Sep;199(9):678-83. doi: 10.1097/NMD.0b013e318229d100. PMID 21878782